CLINICAL TRIAL: NCT06542302
Title: Influence of Various Cervical Sensorimotor Control Challenges on Gait Patterns, Cervical Sensorimotor Control, and Dual-Task Performance During Dynamic Gait-related Tasks
Brief Title: The Effects of Cervical Sensorimotor Control Challenges on Gait Patterns, Cervical Sensorimotor Control During Dynamic Tasks
Status: Not yet recruiting | Type: Observational
Sponsor: National Cheng Kung University (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, YI-JU TSAI, professor, National Cheng Kung University
Other Study IDs: NCKU_Visual Challenge
Record Dates: First submitted 2024-06-19; First posted 2024-08-07 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Neck Pain; Sensorimotor; Gait
Keywords: Sensorimotor control; Chronic neck pain; Oculomotor control; Gait; Balance
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic neck pain group: Pain was unilateral or bilateral between the superior nuchal line and 1st thoracic vertebra; Neck pain persisting for 3 months and above; Average pain intensity of last pain episode was between 2 and 8 based on the numerical rating scale (NRS).
- Asymptomatic adult group: Do not have any complaints of current pain and impairments of neuromusculoskeletal systems within the last 6 months.

SUMMARY:
To investigate the influence of cervical SMC challenges during gait-related dynamic tasks on all task performance and symptoms in patients with CNP.

DETAILED DESCRIPTION:
The goal of this observational study is to learn about the immediate effects of cervical sensorimotor challenges during gait-related dynamic tasks on all task performance and symptoms in patients with CNP .

The main question it aims to answer is:

Does adding sensorimotor challenges in chronic neck pain patient will affect balance and gait performance?

ELIGIBILITY:
Inclusion Criteria:

* Healthy asymptomatic adults will not have any complaints of current pain and impairments of neuromusculoskeletal systems within the last 6 months.
* For patients with CNP

  * Pain was unilateral or bilateral between the superior nuchal line and 1st thoracic vertebra
  * Neck pain persisting for 3 months and above
  * Average pain intensity of last pain episode was between 2 and 8 based on the numeric rating scale (NRS).

Exclusion criteria:

◾For patients with CNP and healthy asymptomatic adults

* Acute or the first onset of neck pain
* Traumatic cause of pain
* Previous fracture or surgery of the spine
* Diagnosed cardiopulmonary diseases, for example, chronic obstructive pulmonary disease, pulmonary tuberculosis, asthma, chronic bronchitis, pulmonary emphysema
* Diagnosed gastrointestinal and abdominal conditions which may interfere daily activities within the past 6 months
* Medical conditions that may affect balance and study procedures (e.g. neurological diseases, vestibular disorders, malignant tumors)
* Metabolic diseases such as anemia and diabetes
* Smoking, plan to pregnant or in pregnancy
* Psychological disorders (affect questionnaire responses)
* Unable to walk independently
* Corrected visual abnormalities or individuals unable to wear contact lenses for vision correction due to the potential interference of wearing VR head-mounted display with glasses.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with chronic neck pain are: (1) pain was unilateral or bilateral between the superior nuchal line and 1st thoracic vertebra, (2) neck pain persisting for 3 months and above, and (3) average pain intensity of last pain episode was between 2 and 8 based on the numeric rating scale (NRS).
Sampling Method: Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Spatiotemporal parameter | One day
  Gait speed (meter/second)
Spatiotemporal parameter | One day
  cadence (steps/minute)
Spatiotemporal parameter | One day
  stride length (meter)
Spatiotemporal parameter | One day
  stride duration (second)
Spatiotemporal parameter | One day
  stance duration (second)
Spatiotemporal parameter | One day
  swing duration (second)
Spatiotemporal parameter | One day
  stance length (meter)
Spatiotemporal parameter | One day
  swing length (meter)
Spatiotemporal parameter | One day
  step width (meter)
Head and Cervical Kinematics | One day
  Mean, range, maximum, and minimum of the angular displacements (degree)
Head and Cervical Kinematics | One day
  Mean and peak angular velocity (m/s) and acceleration (m/^2)
Lower Extremity Kinematics and Kinetics | One day
  Maximum, minimum, and range angular displacement (degree of joint angle)
Lower Extremity Kinematics and Kinetics | One day
  Mean and peak angular velocity and acceleration (m/^2)
Enter of Mass and Center of Pressure (COM-COP) | One day
  A 15-component link-segment model will be used to estimate the location of the total body COM. The center of pressure (COP) data will be derived from the outputs of the AMTI force platform.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No